CLINICAL TRIAL: NCT04010513
Title: A Pilot to Determine the Feasibility of a Hypnosis Intervention for the Treatment of Bladder Pain Syndrome / Interstitial Cystitis
Brief Title: Hypnosis for Bladder Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 832895
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Bladder Pain Syndrome; Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Hypnosis; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental)
  Interventions: Behavioral: Hypnosis
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Hypnosis — Women in the hypnosis group will undergo treatment with three in-person hypnosis sessions and will be given access to hypnosis web-app for at home practice.
  Arms: Hypnosis
Other: Standard of Care — Women in the usual care group will continue their usual care for BPS/IC as dictated by their physicians.
  Arms: Standard of Care

SUMMARY:
This is a pilot randomized control trial of 30 women with interstitial cystitis/bladder pain syndrome to determine the feasibility of delivering a hypnosis intervention or usual care on bladder pain (primary outcome) and cerebral blood flow (secondary outcome). Women in the hypnosis group will undergo treatment with three hypnotherapy sessions in addition to a mobile web-based hypnosis application. Neuroimagning (fMRI) will occur after the first follow up visit.

DETAILED DESCRIPTION:
Available treatments do not provide adequate relief for bladder pain syndrome/interstitial cystitis (BPS/IC), a chronic painful condition that affects 10 million women in the United States. The investigators plan to conduct a pilot randomized control study to determine the feasibility of conducting a combined CBT-hypnosis intervention vs. usual care in women with BPS/IC for a subgroup of women, we will determine the effect of specific hypnotic words on brain function using functional brain imaging. All women will have a pre-existing diagnosis of BPS/IC and their baseline pain prior to therapy and novel (arterial spin labeling) and more traditional (BOLD fMRI) neuroimaging techniques will be collected. Women in the hypnosis group will undergo treatment with three in-person hypnotherapy sessions in addition to a mobile web-based hypnosis application. Women in the usual care group will continue their usual care for BPS/IC. Subjects in both groups will complete a variety of questionnaires on bladder pain, urinary symptoms, sleep, mood, affect, disability, and sexual function before and after treatment. The first follow up visit will occur at the end of treatment (4 weeks after randomization). A select group of patients who are eligible to undergo neuroimaging will be invited to participate in neuroimaging after the first follow up visit. Data will also be collected at a second follow up visit at 2 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Women greater than or equal to 18 years old who are diagnosed with interstitial cystitis or bladder pain syndrome.
* Meet AUA criteria for BPS/IC: an unpleasant sensation (pain, pressure, discomfort) perceived to be related to the urinary bladder, associated with lower urinary tract symptoms of more than six weeks, in the absence of infection or other identifiable causes. - A minimum score greater than or equal to 8 on the Interstitial Cystitis Symptom Index and Problem Index will be required for participation.
* A negative urinalysis or urine culture within 2 months,
* Fluent in English language,
* No changes in IC treatment regimen within 4 weeks of beginning assigned intervention.

Exclusion Criteria:

* Patients who are treatment naive or undergoing 3rd line or higher treatments,
* Pregnant or lactating,
* Unevaluated hematuria, urinary retention,
* A history of cystectomy, urinary diversion or augmentation cystoplasty,
* Other sources of bladder pain (stone, uncontrolled recurrent UTI, radiation cystitis, bladder cancer) or who have a primary diagnosis of another chronic pain condition (such as back pain, fibromyalgia).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female recruitment only
Enrollment: 31 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Improvement in bladder pain self-efficacy as measured by the Female Genitourinary Pain Index | 3 months
  This index is a well validated and widely used instrument for measuring pain in women with BPS/IC

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided